CLINICAL TRIAL: NCT04087447
Title: Vocal and Swallowing Dysfunction Following Thyroid Surgery
Brief Title: Dysfunction Following Thyroid Surgery
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Aya Esam Sharkawy, resident doctor, Assiut University
Other Study IDs: Phoniatrics unit 1/2019
Record Dates: First submitted 2019-09-11; First posted 2019-09-12 (Actual); Last update posted 2019-09-12 (Actual); Status verified 2019-09

CONDITIONS: Thyroidectomy
MeSH Terms: interventions — Thyroidectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Thyroidectomy group: patient undergoing thyroidectomy for simple nodular goiter
  Interventions: Procedure: Thyroidectomy

INTERVENTIONS:
Procedure: Thyroidectomy — Thyroidectomy

SUMMARY:
Voice plays a crucial role in human communication and function. Voice production is multidimensional, involving physiologic, biomechanical, and aerodynamic mechanisms that produce an acoustic output that is perceived by the auditory system. So its important to evaluate patients with voice disorders, whenever possible, to characterize the impact of the disorder(s) on all of the pertinent mechanisms/dimensions.

DETAILED DESCRIPTION:
Voice changes due to laryngeal dysfunction after thyroid surgery are very common complication. However, very few data in the literatures are available which highlights the impact of thyroidectomy and effects of factors, such as patient age, sex, operation type, surgeons experience, laryngeal nerve injury and orotracheal intubation on voice of patients undergoing thyroid surgery. Prabhat AK et al. 2018 reported that, In majority of cases voice changes are transient. The voice recovery time ranges from less than one-month up to 6 months in majority of cases. Transient voice changes, such as voice fatique, and voice weakness or dysphonia are more common and can happen in most of the cases. The transient voice changes usually occurs because one or more of the nerves are irritated either by moving them out of the way during the dissection of thyroid gland or because of the inflammation or oedema that happens after the thyroid surgery.

One of the indices of success in thyroid surgery is the frequency of complications. The most frequent postoperative complications following thyroidectomy are hypocalcemia and airway complications. These are life threatening and have a significant impact on quality of life . Airway complications may result from postoperative haematoma, vocal cord paralysis, laryngeal oedema, and tracheomalacia .

Recurrent laryngeal nerve palsy (RLNP) is a rare but potentially catastrophic complication of thyroid surgery. Damage to a recurrent laryngeal nerve (RLN) with resultant paralysis of the sole abducting muscle (posterior cricoarytenoid) of the vocal folds can cause symptoms ranging from hoarseness in unilateral lesions to stridor and acute airway obstruction in bilateral damage. RLNP following thyroid surgery is one of the leading reasons for medico-legal litigation against surgeons .

Injury of the laryngeal nerves may not be the only cause of voice changes. Other possible causes include injury of the prethyroid strap muscles and cricothyroid muscles or impairment of laryngotracheal movement due to wound contracture after surgical trauma of the soft tissues. A delicate surgical technique may prevent such complications, but it remains to be clarified whether voice alterations may occur after thyroidectomy without any laryngeal nerve injury. Computerized acoustic analysis of the patients undergoing thyroidectomy without laryngeal nerve injury may help determine possible voice changes objectively .

Dysphagia is a typical symptom experinced preoperatively by patients with enlarged thyroid due to a direct compression of the swallowing organs. In these patients, uncomplicated thyroidectomy often leads to improvements in perceptions of swallowing function. However impaired swallowing and neck strangling frequently occur postoperatively. Intraoperative nerve injury regularly causes postoperative dysphagia, but dysphagia is also complained of after uncomplicated thyroidectomies. These symptoms are usually dismissed by the clinicians or attributed to orotracheal intubation. In many patients, correlations for these swallowing disorders cannot be found in objective test results. Reasons for dysphagia and esophageal motility changes after uncomplicated thyroidectomy could be injury of the perithyroidal neural plexus, changes in the laryngeal vascular supply, postoperative adhesions, decreased pressure of the upper esophageal sphincter, or changed position after thyroidectomy .

Investigate non neurogenic causes of vocal and swallowing changes following thyroid surgery: Vocal cord immobility (VCI) is defined as various spectrum of motion impairment in the vocal cord. Although hoarseness is the main symptom in VCI, dysphonia, odynophonia, dysphagia, chronic cough, and laryngospasm can also occur. Visual inspection by a laryngoscopy and electrophysiologic study, such as laryngeal electromyography (LEMG) can help to differentiate the neurogenic and non-neurogenic causes of VCI. The LEMG technique was first introduced by Weddel et al., and needle electrode insertion in small muscles of larynx with assistance of laryngoscopy or in-surgery was first reported in 1950s, followed by the standardized percutaneous electrode insertion technique. LEMG is not only helpful in diagnosing neuromuscular disorder in the larynx, but it can also be used in botulinum toxin or hyaluronic acid injection in vocal cord. In the process of first diagnosing VCI, various systemic diseases can be suspected from the symptoms. Viral or bacterial infections can attribute to post-infectious neuropathies and a wide spectrum of malignancies or tumors present as a paralysis. Also, VCI can be seen in systematic neurologic diseases such as myasthenia gravis, Charcot-Marie-Tooth disease, and multiple sclerosis. With LEMG results, it aids to select other diagnostic tests and determine timing and type of treatments. Furthermore, LEMG results are useful in predicting negative outcomes and their findings can alter definitive treatments. It is important to diagnose VCI of neurogenic causes and to affect treatment and prognosis. However, there are few research studies regarding the association between the clinical characteristics in VCI and LEMG results .

ELIGIBILITY:
Inclusion Criteria:

* benign and malignant thyroid disease normal voice controlled thyroid hormones level

Exclusion Criteria:

* Age below 18 years any cardiac, renal,hepatic, respiratory, mental can interfere with the surgery any voice changes due to any cause before surgery previous head and neck surgery neurological dysfunctions

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adults patients undergoing thyroid surgery
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-01-01 (Estimated); Primary Completion 2021-01-01 (Estimated); Study Completion 2021-07-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of voice function | from end of surgery till two months after surgery
  fibroptic endoscopic assessment of voice function
Assessment of swallowing function | from end of surgery till two months after surgery
  fibroptic endoscopic assessment of swallowing function

SECONDARY OUTCOMES:
postoperative care of these patients | from end of surgery till two months after surgery
  this includes improve voice and swallowing dysfunction

IPD SHARING:
Plan to Share IPD: Undecided